CLINICAL TRIAL: NCT01967056
Title: Predictors of Respiratory Failure Following Extubation in Teh Surgical Intensive Care Unit (SICU)
Brief Title: Predictors of Respiratory Failure Following Extubation in the SICU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Ulrich Schmidt, Associate Professor of Anesthesia, Massachusetts General Hospital
Other Study IDs: 2012P001783
Record Dates: First submitted 2013-10-16; First posted 2013-10-22 (Estimated); Last update posted 2013-10-22 (Estimated); Status verified 2013-10

CONDITIONS: Muscle Weakness; Renal Failure; Respiratory Comorbidities
Keywords: Muscle strength; respiratory failure; extubation failure; intensive care unit; outcome prediction
MeSH Terms: conditions — Muscle Weakness; Renal Insufficiency; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Respiratory failure following extubation causes significant morbidity and increases mortality in teh surgical intensive care unit (SICU). However the causes of respiratory failure following extubation remain poorly understood. The investigators hypothesize that extubation failure can be predicted based on preoperative risk factors as well as ICU acquired morbidities including muscle weakness and renal failure.

DETAILED DESCRIPTION:
Both extubation delay and extubation failure are related to adverse outcomes. A spontaneous breathing trial is therefore recommended to predict extubation readiness. However, depending on the disease entity and local culture, a range of 10-20 per cent incidence of extubation failure has been described from tertiary care hospitals. The aim of this trial is to identify additional variables in surgical patients that can be used to support a clinician's decision on whether or not to extubate a patient's trachea.

Te investigators have recently developed and validated the SPORC (Brueckmann, 2013), a score that predicts the risk of extubation failure following surgery based on patients comorbidities and the acuity of the disease leading to surgery, and the investigators hypothesize that the SPORC will also predict extubation failure in the surgical ICU.

In addition, it is likely that ICU acquired morbidity also predicts extubation failure. In fact, the investigators have recently shown that muscle weakness is a predictor of aspiration (Mirzakhani, 2013), and the investigators speculated that muscle weakness may also respiratory failure after extubation.

Finally, it has been suggested that the increased mortality seen in patients with acute kidney injury (AKI) requiring continuous renal replacement therapy (CRRT) versus end stage renal disease (ESRD) patients requiring CRRT can be attributed to an increased need for mechanical ventilation. (Walcher, 2011). Therefore, the investigators also hypothesize that acute kidney injury increases the vulnerability of patients to postextubation respiratory failure.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years of age or greater)
* Patients who have been extubated following mechanical ventilation in the surgical ICU

Exclusion Criteria:

* Preexisting end-stage renal disease
* Neurological disorder associated with severe muscle weakness
* Goals of care focused on comfort

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of patients used for this study will be those admitted to the Surgical Intensive Care Unit
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-06 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Respiratory Failure | 30 days
  The investigators defined respiratory failure as a composite endpoint including reintubation within 72 hours, use of non-invasive ventilation for treatment of extubation failure, and tracheostomy during hospitalization (expected time of 30 days post extubation)

SECONDARY OUTCOMES:
Reintubation within 72 hours | 72 hours
  The investigators will follow patients and observe whether they require reintubation within 72 h
Non-invasive ventilation for treatment of extubation failure | 72 hours
  The investigators will follow patients and observe whether they require non-invasive ventilation for extubation failure
Tracheostomy | Patients will be followed for 30 days of hospitalization
SICU length of stay | 180 days
Hospital length of stay | 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Schmidt, MD, Principal Investigator — The Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Brueckmann B, Villa-Uribe JL, Bateman BT, Grosse-Sundrup M, Hess DR, Schlett CL, Eikermann M. Development and validation of a score for prediction of postoperative respiratory complications. Anesthesiology. 2013 Jun;118(6):1276-85. doi: 10.1097/ALN.0b013e318293065c. PMID 23571640
- [Background] Mirzakhani H, Williams JN, Mello J, Joseph S, Meyer MJ, Waak K, Schmidt U, Kelly E, Eikermann M. Muscle weakness predicts pharyngeal dysfunction and symptomatic aspiration in long-term ventilated patients. Anesthesiology. 2013 Aug;119(2):389-97. doi: 10.1097/ALN.0b013e31829373fe. PMID 23584384
- [Background] Walcher A, Faubel S, Keniston A, Dennen P. In critically ill patients requiring CRRT, AKI is associated with increased respiratory failure and death versus ESRD. Ren Fail. 2011;33(10):935-42. doi: 10.3109/0886022X.2011.615964. Epub 2011 Sep 13. PMID 21910664
- [Background] Bittner EA, Schmidt UH. Tracheal reintubation: caused by "too much of a good thing"? Respir Care. 2012 Oct;57(10):1687-91. doi: 10.4187/respcare.02082. No abstract available. PMID 23013905
- [Derived] Fuchs G, Thevathasan T, Chretien YR, Mario J, Piriyapatsom A, Schmidt U, Eikermann M, Fintelmann FJ. Lumbar skeletal muscle index derived from routine computed tomography exams predict adverse post-extubation outcomes in critically ill patients. J Crit Care. 2018 Apr;44:117-123. doi: 10.1016/j.jcrc.2017.10.033. Epub 2017 Oct 23. PMID 29096229
- [Derived] Piriyapatsom A, Williams EC, Waak K, Ladha KS, Eikermann M, Schmidt UH. Prospective Observational Study of Predictors of Re-Intubation Following Extubation in the Surgical ICU. Respir Care. 2016 Mar;61(3):306-15. doi: 10.4187/respcare.04269. Epub 2015 Nov 10. PMID 26556899